CLINICAL TRIAL: NCT02595996
Title: An Intra-patient Dose Escalation Study of Propranolol in Patients With Lymphedema
Brief Title: Propranolol Dose Escalation in Lymphedema in Patients
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of funding
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, June Wu, Assistant Professor of Surgery, Columbia University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AAAP9262
Record Dates: First submitted 2015-09-18; First posted 2015-11-04 (Estimated); Results first posted 2021-10-22 (Actual); Last update posted 2021-10-22 (Actual); Status verified 2021-09

CONDITIONS: Primary Lymphedema
MeSH Terms: conditions — Lymphedema | interventions — Propranolol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (Experimental): Patients will be given propranolol in escalating doses
  Interventions: Drug: Propranolol

INTERVENTIONS:
Drug: Propranolol — escalating doses of propranolol from 1mg/kg/day to 2mg/kg/day to 3mg/kg/day
  Other Names: Inderal

SUMMARY:
This is a study to investigate the safety and efficacy of propranolol in the treatment of patients with primary lymphedema. The primary goal is to assess patient tolerability of increasing doses of propranolol. The secondary goal is to assess lymphedema symptoms and signs in response to propranolol treatment.

DETAILED DESCRIPTION:
Lymphatic malformations (LMs) arise from abnormal development of lymphatic vasculature. Primary lymphedema is considered a form of LM. Recently, results in the investigators' laboratory demonstrated that propranolol, a pan beta-adrenergic receptor (βAR) antagonist, had cytotoxic and anti-proliferative effects against cells isolated from LM tissues. Preliminary results from treating symptomatic LM patients with propranolol at a dose range from 0.7-1mg/kg/day demonstrated a 70% positive response rate, with patients reporting improvement in their symptoms.

Propranolol has been used for different indications for many years. Propranolol is accepted for use in infants with hemangiomas and supraventricular tachycardia. Hemangeol was approved by the FDA for use in infants with hemangiomas. However, βAR antagonists are not without potential adverse effects, including hypotension, bradycardia, hypoglycemia, bronchospasms, and sleep disturbances. FDA-approved dose range for treating hemangiomas in infants (>5 weeks old, >2kg) ranged from 1-3mg/kg/day in divided doses. Propranolol doses of up to 4mg/kg/day has been used for pediatric supraventricular tachycardia. Therefore, the investigator's experience with propranolol use in LM patients have been at the low end of most accepted clinical indications. The investigators propose to escalate propranolol dosages up to 3mg/kg/day in this study, well below the dose ranges currently used in clinical settings.

This dose range of 0.7-1mg/kg/day was chosen for LM patients as it was the low end of dose range for infants treated with propranolol for problematic hemangiomas, a related vascular anomaly. At this dose, no significant hemodynamic adverse effects were noted in LM patients. However, when patients stopped propranolol or their dose fell below 0.7mg/kg/day, they suffered rebound worsening of their symptoms. Moreover, inflammatory events such as infections temporarily overcame the effects of 0.7-1mg/kg/day of propranolol. Thus, it is unknown whether maximum propranolol efficacy was achieved at the current dose range. The investigators propose to examine whether optimized propranolol usage for treatment of LM patients has been achieved. The primary endpoint for this study is to ascertain whether LM patients can tolerate higher doses of propranolol, as measured by known propranolol adverse effects and patient-reported symptoms. A secondary endpoint will address whether patient-reported LM symptoms and quality of life are improved with higher doses of propranolol; objective findings such as LM size on physical examination and imaging studies will be analyzed as well. In addition, LM tissue biopsies will acquired from patients before and after propranolol treatment for further analyses of disease progression.

ELIGIBILITY:
Inclusion Criteria:

* Primary lymphedema
* Measurable disease
* Adequate functional status: Karnofsky >50% (>age 16), Lanky >50 (<age 16),
* No prior therapy within 4 weeks of enrollment
* Adequate bone marrow, renal function, cardiac, and pulmonary function, negative pregnancy test (for women).

Exclusion Criteria:

* Secondary lymphedema
* Patients already receiving other investigational drugs
* Patients with known contraindications to receiving propranolol
* Other medical comorbidities including but not limited to: pheochromocytoma, bradycardia, bronchospasm/reactive airway disease, decompensated heart failure, heart block, ongoing active infections.

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2017-06-07 (Actual); Primary Completion 2020-10-08 (Actual); Study Completion 2020-10-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: June K. Wu, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 1
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients That Tolerated Propranolol
Description: To assess whether patients tolerated propranolol
Time Frame: 8 weeks
Population: Study terminated due to lack of funding. Data was not analyzed or disclosed due to subject confidentiality being an issue (n=1).
Arm/Group | Treatment
Number analyzed (Participants) | 0

2. Secondary Outcome: Number of Patients With Improved Quality of Life Based on Self-reported Questionnaires
Description: To assess subjective lymphedema symptoms improvements only - whether patients' general quality of life symptoms improved on propranolol treatment by self-reported questionnaires (SF 36)
Time Frame: 8 weeks
Population: as for outcome 1
Arm/Group | Treatment
Number analyzed (Participants) | 0

3. Secondary Outcome: Number of Patients With Decreased Fluid Retention by Weight
Description: To assess whether patients' lymphedema signs are improved on propranolol by weight (BMI kg/m^2) - objective signs of improvement of their lymphedema
Time Frame: 8 weeks
Population: as for outcome 1
Arm/Group | Treatment
Number analyzed (Participants) | 0

4. Secondary Outcome: Number of Patients With Lower Limb Discrepancy
Description: To assess whether patients' lymphedema signs are improved on propranolol by limb girth discrepancy measurement (%) - objective signs of improvement of their lymphedema
Time Frame: 8 weeks
Population: as for outcome 1
Arm/Group | Treatment
Number analyzed (Participants) | 0

5. Secondary Outcome: Number of Patients With Decreased Fluid Retention on MRI
Description: To assess whether patients' lymphedema signs are improved on propranolol - the decrease in fluid retention will be calculated by the measurement of fat (a number) divide by the measurement of fluid (a number) to yield a ratio - if a patient has a lower ratio at 8 weeks than at baseline, they will be reported in this category.
Time Frame: baseline to 8 weeks
Population: as for outcome 1
Arm/Group | Treatment
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Up to 8 weeks
Arm/Group | Treatment
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 0/1

LIMITATIONS AND CAVEATS:
Study terminated due to lack of funding. Data was not analyzed or disclosed due to subject confidentiality being an issue (n=1).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-22): https://cdn.clinicaltrials.gov/large-docs/96/NCT02595996/Prot_SAP_000.pdf